CLINICAL TRIAL: NCT02388438
Title: Efficiency and Safety of Demineralized Bone Matrix in the Proximal Opening Wedge Osteotomy for Hallux Valgus Deformity
Brief Title: Demineralized Bone Matrix in Opening Wedge Osteotomy for Hallux Valgus Deformity
Acronym: DBM
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Severance Hospital (Other)
Responsible Party: Principal Investigator, Woojin Choi, Orthopedic part, Severance Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SS-13-Bongener; CGBIOB1306 (Other Grant/Funding Number: CGBIO CO., LTD.)
Record Dates: First submitted 2015-03-04; First posted 2015-03-17 (Estimated); Last update posted 2015-03-17 (Estimated); Status verified 2015-03

CONDITIONS: Hallux Valgus
Keywords: demineralized bone matrix
MeSH Terms: conditions — Hallux Valgus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Demineralized bone matrix (Experimental): Applied demineralized bone matrix when investigator conduct hallux valgus surgery.
  Interventions: Device: Bongener

INTERVENTIONS:
Device: Bongener

SUMMARY:
This study evaluates the demineralized bone matrix in "Hallux valgus".

DETAILED DESCRIPTION:
Demineralized bone matrix use for filling in the space removed bone in open wedge osteotomy and correction. The purpose this study is to test therapeutic benefits of demineralized bone matrix.

Investigator will recruit thirty patients. Total evaluation period will be 12 months. In this period, investigator will examine correction rate, fusion rate, functional test, adverse event.

ELIGIBILITY:
Inclusion Criteria:

* (1) The patient ranging in age from 20 to 75 years
* (2) Has to be operated over 5mm osteotomy for correcting hallux valgus.
* (3) The patients who were able to comply with the research protocol.

Exclusion Criteria:

* (1) Bursitis in metatarsal bones has affected surgery.
* (2) Has rheumatism
* (3) The patient who has clinical sign of infection on the operated site at pre-screening
* (4) Patient who has failure of peripheral blood circulation caused by chronic disease and neurological symptoms
* (5) In the opinion of investigator, the patient is not suitable to participate in this study

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-04; Primary Completion 2014-08 (Actual); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
days to union from applied demineralized bone matrix | up to 12months
  Examine the days from applied medical device to union.

SECONDARY OUTCOMES:
Complete fusion rate after applied medical device. | up to 12months
  Examine the fusion rate of osteotomy site and evaluate fusion rate according to definition of protocol with every visit.
Complete correction rate after applied medical device. | up to 12months
  Examine the corrected degree of hallux valgus and evaluate correction rate according to definition of protocol with every visit
Change from baseline AOFAS(American Orthopaedic Foot and Ankle Society) at 12 months. | change form baseline at 12months
  Evaluate the AOFAS with every visit. Compared the AOFAS score with baseline AOFAS score.

OTHER OUTCOMES:
Adverse events | up to 12months
  Evaluate adverse event after applied medical device. Examine adverse every visit.